CLINICAL TRIAL: NCT04527406
Title: Early Hemivertebra Resection of Congenital Hemivertebra in Very Young Children: A Randomized Clinical Study
Brief Title: Early Surgical Intervention of Congenital Hemivertebra in Young Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEMI 1.1
Record Dates: First submitted 2020-08-24; First posted 2020-08-26 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Congenital Hemivertebra
Keywords: Congenital hemivertebra; Young Children; posterior hemivertebra resection

STUDY DESIGN:
Intervention Model Description: The research subjects are randomly assigned to the early surgery group (experimental group) or traditional surgery group (control group) at a ratio of 1:1
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor conduct independent statistical analysis and evaluation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early surgical group (Experimental): The subjects in this group received early surgical treatment, and they are arranged to be admitted to the hospital for surgical treatment after admission. The operation choice is posterior hemivertebrae resection + posterior pedicle screw placement + scoliosis correction.
  Interventions: Procedure: posterior hemivertebra resection
- Traditional surgical treatment (Active Comparator): This group of subjects received conservative treatment with custom-made braces to delay the progression of scoliosis. It is planned to use the classic posterior hemivertebrae resection + posterior pedicle screw placement + scoliosis correction to complete the correction around the age of 5.
  Interventions: Procedure: conservative treatment+ delayed posterior hemivertebra resection

INTERVENTIONS:
Procedure: posterior hemivertebra resection — The subjects in early surgical group are arranged to be admitted to for surgical treatment very soon. The operation choice is posterior hemivertebrae resection + posterior pedicle screw placement + scoliosis correction. During operation pedicle screws are placed in the adjacent vertebrae of the head and tail of the Hemivertebra. Wedge resection of the hemivertebrae is performed afterward. Finally, two rods are placed between the pedicle screws. Intraoperative fluoroscopy confirms that the internal fixation position is good.
  Arms: Early surgical group
Procedure: conservative treatment+ delayed posterior hemivertebra resection — In traditional surgical group, subjects received conservative treatment firstly with custom-made braces to delay the progression of scoliosis. It is planned to use the classic posterior hemivertebrae resection + posterior pedicle screw placement + scoliosis correction to complete the correction around the age of 5. The operation choice is identical with early surgical group. During operation pedicle screws are placed in the adjacent vertebrae of the head and tail of the Hemivertebra. Wedge resection of the hemivertebrae is performed afterward. Finally, two rods are placed between the pedicle screws. Intraoperative fluoroscopy confirms that the internal fixation position is good.
  Arms: Traditional surgical treatment

SUMMARY:
Early treatment of congenital hemivertebrae is very important. The investigators design this study to figure out how early hemivertebrae resection be apply to children. Children aged 3-5 years old diagnosed as congenital hemivertebrae will be randomly divided into early operation group and control group. The early operation group will undergo posterior hemivertebra resection. The control group received brace plaster fixation to reduce the progression of scoliosis, and then will undergo operation after 5 years old. Primary Outcome Measure is the length of spine surgery.

DETAILED DESCRIPTION:
Early diagnosis and early effective treatment of congenital hemivertebrae can correct the deformities.Therefore, traditionally, children with a clear diagnosis should be fixed with a brace to delay the aggravation of scoliosis and then undergo surgery after 5 years of age. The design of this study is to conduct a single-center randomized controlled study. Children aged 3-5 years old diagnosed as congenital hemivertebrae will be randomly divided into the early operation group and the control group. The early operation group will undergo posterior hemivertebra resection. The control group received brace plaster fixation to reduce the progression of scoliosis, and posterior scoliosis correction will be performed after the age was over 5 years old. The primary outcome measures are the length of spine surgery for the two groups of children. The secondary outcome measures are change of scoliosis cobb angle, by comparing preoperative and postoperative cobb angle changes. It is expected that the early treatment group will shorten the length of surgery due to the smaller degree of scoliosis. Our research is expected to broaden the age-adaptation of classic spinal surgery in the field of pediatric spine.

ELIGIBILITY:
Inclusion Criteria:

* Single-segment thoracic or lumbar hemivertebrae scoliosis diagnosed by X-ray and CT.

Exclusion Criteria:

* Diagnosed with syndrome of scoliosis, osteochondrodysplasia, multi-segment hemivertebrae deformity, cervical hemivertebrae deformity

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Duration of surgery | The operation time： from the beginning of the surgical skinning to the end of the surgical suture
  The length of posterior hemivertebra resection operation time, acquired in the operation record from hospital

SECONDARY OUTCOMES:
change of scoliosis cobb angle | intraoperative
  X-ray measurement of scoliosis cobb angle, by compare the preoperative and postoperative cobb angle changes to obtain the degree of scoliosis correction

CONTACTS AND LOCATIONS:
Overall Officials: Dahui Wang, MD-PhD, Principal Investigator — Children's hospital of fudan uviversity, shanghai, China

IPD SHARING:
Plan to Share IPD: No
depend on correspond

REFERENCES:
- [Background] Ginsburg G, Mulconrey DS, Browdy J. Transpedicular hemiepiphysiodesis and posterior instrumentation as a treatment for congenital scoliosis. J Pediatr Orthop. 2007 Jun;27(4):387-91. doi: 10.1097/01.bpb.0000271312.95621.b0. PMID 17513957